CLINICAL TRIAL: NCT06024226
Title: Role of Myeloid Derived Suppressive Cells (MDSCs) and Cancer Stem Cells and Their Cross Talks in Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Role of MDSCs and Cancer Stem Cells and Their Cross Talks in NSCLC
Acronym: MyéloLungSC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/35
Record Dates: First submitted 2023-08-28; First posted 2023-09-06 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Lung Neoplasms; Myeloid-Derived Suppressor Cells; Immunosuppression
Keywords: Lung cancer; Immunosuppression; Immuno-oncology; Antitumor immune escape; Invasion
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with lung carcinoma surgically treated by surgery only
  Interventions: Procedure: Tumor samples

INTERVENTIONS:
Procedure: Tumor samples — Tumor samples will be collected by the pathologist at the reception of the tumor removed during surgery

SUMMARY:
Immunotherapy have revolutionized the field of oncology, but response rates are low and all patients relapse, due to cellular and soluble immunosuppressive mechanisms. MDSC are one of the most important immunosuppressive cells, that also harbour non immunologic functions, favouring cancer invasion. These non immunologic functions of MDSC in lung cancer will be better characterized. Indeed, cellular mechanisms will be analysed by in vitro studies, assessing the effect of immunosuppressive cells, provided by fresh tumor samples, on phenotype and functions of lung cancer cell lines. The aim of this study is to better characterize immunosuppressive landscape of NSCLC and mechanisms involved in their protumor functions.

DETAILED DESCRIPTION:
In recent years, immune-based therapies have revolutionized the field of oncology by significantly improving survival of cancer patients. Despite sustained responses, only 20% to 40% of cancer patients respond. It has become clear that the immunosuppressive environment induced by tumor through cellular and/or soluble pathways critically contribute to hinder efficient antitumor immunity. The inhibition of these immunosuppressive networks thus represents an essential prerequisite for the improvement of responses to anticancer immunotherapies. Several immune cell populations have been identified as key actors of tumor-induced immunosuppression, among which are myeloid-derived suppressor cells (MDSC) and regulatory T lymphocytes (Treg). However, in non-small cell lung cancers (NSCLC), the prognostic role of these cells, the mechanisms underlying their immunosuppressive functions, their "non-immunological" protumoral functions and their role in dampening the efficacy of immunotherapies in clinical practice are less characterized. The aim of this project is to better characterize the non immunologic functions of MDSC. We propose to assess in vitro the non-immunological pro-tumor functions of MDSC isolated from lung cancer patients

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients
* lung carcinoma surgically treated by surgery only

Exclusion Criteria:

* patient receiving chemotherapy, radiotherapy or immunotherapy in the neoadjuvant setting (all objectives)
* patient with concomitant or previous cancer (in the 2 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung carcinoma surgically treated by surgery only
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Comparative analysis of the modifications of phenotype and functions of lung cancer cell lines when exposed to MDSC extracted from patient tumor tissue | At the time of surgery only, when fresh tumor is resected
  Functional in vitro studies of the effect of MDSC extracted from resected NSCLC prospectively collected on phenotype and function of lung cancer cell lines

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux - Hôpital Saint-André, Service d'Oncologie Médicale, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No